CLINICAL TRIAL: NCT00327353
Title: Single-Centre Randomised Open Crossover Study to Examine the Influence of Different Internal Resistances of Discus and Turbohaler Respectively on the Effects of Salmeterol and Formoterol in Asthmatic Subjects
Brief Title: Influence Of Different Airflow Resistances On Drug Effect Of 50μg Salmeterol And 6 μg Formoterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 101182; TURBOHALER Faktor
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Asthma
Keywords: Asthma; Salmeterol; Formoterol; Airway resistance
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Salmeterol Xinafoate

INTERVENTIONS:
Drug: formoterol (TURBOHALER)
Drug: Salmeterol (DISKUS)
  Other Names: formoterol (TURBOHALER)

SUMMARY:
Effect of inhaled drugs administered as dry powder is not only dependent on drug efficacy but also on technical properties of the inhalers. Different inhalers have different internal resistances and therefore it is expected that patients with limited airflow may have different exposure rates of drugs delivered from different devices

ELIGIBILITY:
Inclusion criteria:

* Asthma Reversibility >15% and 200 ml in total FEV1 <85% of normal

Exclusion criteria:

* Smoking history >20 pack years Treatment with ICS >500μg Fluticasone or aquivalent in the last 4 weeks Asthma exacerbation in the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77
Dates: Start 2004-01

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) under time curve 0.5-6 hours after inhalation of study medication

SECONDARY OUTCOMES:
Airway resistances and peak FEV1 measured 0.5, 1, 2, 4 and 6 hours after inhalation of study drug

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (2):
- Germany (2):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Berlin, State of Berlin